CLINICAL TRIAL: NCT04800523
Title: The "UroMonitor Trial": Safety, Feasibility, and Tolerability of UroMonitor Insertion in Spinal Cord Injury.
Brief Title: "UroMonitor Trial" in Spinal Cord Injury.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar study already completed
Sponsor: University of British Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian Kwon, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H20-01267
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 - Non-functional Device (Experimental): a non-functional UroMonitor will be inserted by urologist.
  Interventions: Device: UroMonitor System

INTERVENTIONS:
Device: UroMonitor System — Implantable device to wirelessly and without catheters monitor the neurogenic bladder on an ambulatory basis

SUMMARY:
This study aims to determine if a non-functioning UroMonitor device can be safely inserted, monitored, and removed in patients with SCI.

DETAILED DESCRIPTION:
This prospective, observational study will be conducted with 10 patients with chronic thoracolumbar SCI who are already undergoing routine UDS studies as part of their care. Following their routine UDS, a non-functioning UroMonitor device will be inserted and removed after 3 hours. Participants' symptoms will be monitored after the UroMonitor is inserted, following the 3 hour monitoring period, and again after UroMonitor removal. A second cystoscopy will be conducted for research purposes after removal to examine the urethra and bladder for any irritation or trauma. During insertion and removal, the urologist will document the time required for insertion and any difficulties encountered

ELIGIBILITY:
Inclusion Criteria:

1. Cervical or Thoracolumbar (T2-L1 spinal level) spinal cord injury with AIS A, B, C, or D severities of injury.
2. Age 17-75.
3. At least 1 year post-injury.
4. At least one prior urodynamics study in the past 12 months that has objectively documented abnormalities on bladder function consistent with an upper motor neuro lesion.
5. History of neurogenic bladder symptoms requiring some form of intervention (e.g. clean intermittent catheterization, condom catheter)

Exclusion Criteria:

1. Lumbar injuries (L2-S1 spinal level) where the injury is primarily to the cauda equina and not to spinal cord.
2. History of autonomic dysreflexia (such individuals are excluded to minimize the chance of inducing autonomic dysreflexia with device insertion).
3. Active urinary tract infection.
4. Past urethral or bladder reconstruction surgery

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Participant Symptoms During Implantation | Day 1 Timepoint: post insertion
  11-point numerical visual analogue scale for the participant to document discomfort during the implantation of the UroMonitor.
Device Insertion Form for Urology Specialist | Day 1 Timepoint: post insertion
  Study form registers the data on application of the device, such as the time and ease of insertion.
Participant Symptoms During 3-Hour Monitoring | Day 1 Timepoint: 1 hr post insertion
  Study form used for the purpose of registering data on details of participant symptoms during the 3-hour monitoring period
Device Removal Form for Urology Specialist | Day 1 Timepoint: post device remove
  Study form used for the purpose of recording the condition of the device and patient's experience at the time of sensor removal
Participant Symptoms during Device Removal Form | Day 1 Timepoint: post device remove
  Data on details of patient symptoms during device removal is recorded with this form
Second Cystoscopy Form for Urology Specialist | Day 1 Timepoint: post secondary cyctoscopy
  This form is used for the purpose of recording the existence of irritation in bladder or urethra after the removal of the device

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kwon, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada